CLINICAL TRIAL: NCT01655706
Title: Integrated Biological Markers for the Prediction of Treatment Response in Depression
Brief Title: Canadian Biomarker Integration Network for Depression Study
Acronym: CAN-BIND-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Toronto (Other); University of Calgary (Other); University of British Columbia (Other); McGill University (Other); Queen's University (Other); Centre for Addiction and Mental Health (Other); McMaster University (Other)
Responsible Party: Principal Investigator, Sidney Kennedy, Psychiatrist, Pricipal Investigator, University Health Network, Toronto
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-0917-A
Record Dates: First submitted 2012-07-27; First posted 2012-08-02 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Major Depressive Disorder
Keywords: major depression; major depressive disorder; biomarkers; escitalopram; aripiprazole; MDD; neuroimaging; proteomic; genomics
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Dexetimide; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- escitalopram (10-20mg) (Active Comparator): Patients are on escitalopram for 8 weeks. At Week 8, patients will be assessed as 'responders' or 'non-responders'. 'Responders' will continue on escitalopram until study endpoint.
  Interventions: Drug: escitalopram
- aripiprazole (2-10mg) (Active Comparator): At Week 8, patients assessed as 'non-responders' will be given aripiprazole as an add-on treatment to escitalopram.
  Interventions: Drug: escitalopram; Drug: aripiprazole

INTERVENTIONS:
Drug: escitalopram — Patients will be given escitalopram for the first 8 weeks of the trial. At week 8, patients who are assessed as 'responders' will continue on escitalopram until study endpoint.
  Other Names: Cipralex
Drug: aripiprazole — At Week 8, patients assessed as 'non-responders' will be given aripiprazole as an add-on treatment to escitalopram.
  Other Names: Abilify
  Arms: aripiprazole (2-10mg)

SUMMARY:
This study is a pilot to assess feasibility of the protocol in patients and controls across six participating sites. The goal is to identify biological markers (biomarkers)that can be measured at baseline or early in treatment to predict treatment outcome in individual patients with Major Depressive Disorder (MDD). Biomarkers of interest will be clinical (using interview and self-report measures), molecular (from blood samples) and neurobiological (using neuroimaging and EEG).

DETAILED DESCRIPTION:
This is a study to collect clinical and biomarker data which will be used to build models to predict treatment response. This is not a study to evaluate efficacy of medications, as medications in this study have been approved by Health Canada and are widely used for the treatment of MDD.

This is an open label study involving MDD patients and healthy controls.Patients with a diagnosis of MDD and a current major depressive episode (MDE) will receive open-label standard of care treatment with escitalopram (10-20mg). Healthy controls will not receive medication; however, they will go through clinical assessments, blood collection and neuroimaging procedures.

At week 8, patients will be assessed for medication response (response is defined as ≥ 50% reduction in MADRS scores from baseline). Responders will continue medication at their effective dose until study endpoint while non-responders will receive open label add-on treatment with aripiprazole (2-10mg).

There are approximately 7 clinic visits over a 16 week period during which patients and healthy controls will undergo clinician administered scales and self reports, provide blood and urine samples (which will undergo proteomic and genomic analyses) as well as neuroimaging (fMRI and EEG).

At the end of the study, mathematical modeling methods will be used to integrate the data from the various modalities to see which features best predict treatment outcome.

ELIGIBILITY:
For Depressed patients:

Inclusion Criteria:

* Outpatients who are 18-60 years of age
* Meet DSM-IV-TR criteria for Major Depressive Episode in Major Depressive Disorder by the MINI
* Episode duration ≥ 3 months
* Free of psychotropic medications for at least 5 half-lives (i.e. 1 week for most antidepressants, 5 weeks for fluoxetine) before baseline Visit 1
* MADRS ≥ 24
* Fluency in English, sufficient to complete the interviews and self-report questionnaires

Exclusion Criteria:

* Any Axis I diagnosis other than MDD that is considered the primary diagnosis
* Bipolar I or Bipolar II diagnosis
* Presence of a significant Axis II diagnosis (borderline, antisocial)
* High suicidal risk, defined by clinician judgment
* Substance dependence/abuse in the past 6 months
* Presence of significant neurological disorders, head trauma or other unstable medical conditions
* Pregnant or breastfeeding
* Failure of 3 or more adequate pharmacologic interventions (as determined by the Antidepressant Treatment History Form)
* Started psychological treatment within the past 3 months with the intent of continuing treatment
* Patients who have previously failed escitalopram or showed intolerance to escitalopram and patients at risk for hypomanic switch (i.e. with a history of antidepressant hypomania)

Inclusion criteria for Healthy Controls:

* 18 to 60 years of age
* No history of Axis I or Axis II disorders, as determined by the MINI.
* Fluency in English, sufficient to complete the interviews and self-report questionnaires.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 211 (Actual)
Dates: Start 2012-04-23 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in MADRS (Montgomery-Asberg Depression Rating Scale) scores from baseline | Week 8, Week 16
  Clinical response (≥ 50% reduction in MADRS scores from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Sidney Kennedy, MD, Principal Investigator — University Health Network, University of Toronto
Locations (6):
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - University Health Network, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
This study is funded by the Ontario Brain Institute (OBI). Data collected from this study is entered into a research database called "Brain-CODE", deployed at a High Performance Computer Virtual Lab (HPCVL). The HPCVL supports the regulatory-compliant (e.g. 21 CRF Part 11, HIPPA, PIPEDA) processes for securing privacy of healthcare data.

REFERENCES:
- [Background] Kennedy SH, Downar J, Evans KR, Feilotter H, Lam RW, MacQueen GM, Milev R, Parikh SV, Rotzinger S, Soares C. The Canadian Biomarker Integration Network in Depression (CAN-BIND): advances in response prediction. Curr Pharm Des. 2012;18(36):5976-89. doi: 10.2174/138161212803523635. PMID 22681173
- [Background] Lam RW, Milev R, Rotzinger S, Andreazza AC, Blier P, Brenner C, Daskalakis ZJ, Dharsee M, Downar J, Evans KR, Farzan F, Foster JA, Frey BN, Geraci J, Giacobbe P, Feilotter HE, Hall GB, Harkness KL, Hassel S, Ismail Z, Leri F, Liotti M, MacQueen GM, McAndrews MP, Minuzzi L, Muller DJ, Parikh SV, Placenza FM, Quilty LC, Ravindran AV, Salomons TV, Soares CN, Strother SC, Turecki G, Vaccarino AL, Vila-Rodriguez F, Kennedy SH; CAN-BIND Investigator Team. Discovering biomarkers for antidepressant response: protocol from the Canadian biomarker integration network in depression (CAN-BIND) and clinical characteristics of the first patient cohort. BMC Psychiatry. 2016 Apr 16;16:105. doi: 10.1186/s12888-016-0785-x. PMID 27084692
- [Derived] Mazurka R, Cunningham S, Hassel S, Foster JA, Nogovitsyn N, Fiori LM, Strother SC, Arnott SR, Frey BN, Lam RW, MacQueen GM, Milev RV, Rotzinger S, Turecki G, Kennedy SH, Harkness KL. Relation of hippocampal volume and SGK1 gene expression to treatment remission in major depression is moderated by childhood maltreatment: A CAN-BIND-1 report. Eur Neuropsychopharmacol. 2024 Jan;78:71-80. doi: 10.1016/j.euroneuro.2023.12.003. Epub 2023 Dec 20. PMID 38128154
- [Derived] Phaterpekar T, Nunez JJ, Morton E, Liu YS, Cao B, Frey BN, Milev RV, Muller DJ, Rotzinger S, Soares CN, Taylor VH, Uher R, Kennedy SH, Lam RW. Machine Learning Prediction of Quality of Life Improvement During Antidepressant Treatment of Patients With Major Depressive Disorder: A STAR*D and CAN-BIND-1 Report. J Clin Psychiatry. 2023 Nov 15;85(1):23m14864. doi: 10.4088/JCP.23m14864. PMID 37967350
- [Derived] Islam F, Magarbeh L, Elsheikh SSM, Kloiber S, Espinola CW, Bhat V, Frey BN, Milev R, Soares CN, Parikh SV, Placenza F, Hassel S, Taylor VH, Leri F, Blier P, Uher R, Farzan F, Lam RW, Turecki G, Foster JA, Rotzinger S, Kennedy SH, Muller DJ. Influence of CYP2C19, CYP2D6, and ABCB1 Gene Variants and Serum Levels of Escitalopram and Aripiprazole on Treatment-Emergent Sexual Dysfunction: A Canadian Biomarker Integration Network in Depression 1 (CAN-BIND 1) Study. Can J Psychiatry. 2024 Mar;69(3):183-195. doi: 10.1177/07067437231203433. Epub 2023 Oct 5. PMID 37796764
- [Derived] Espinola CW, Khoo Y, Parmar R, Demchenko I, Frey BN, Milev RV, Ravindran AV, Parikh SV, Ho K, Rotzinger S, Lou W, Lam RW, Kennedy SH, Bhat V. Males and females differ in reported sexual functioning with escitalopram treatment for major depressive disorder: A CAN-BIND-1 study report. J Psychopharmacol. 2022 May;36(5):604-613. doi: 10.1177/02698811221095832. Epub 2022 May 12. PMID 35546043
- [Derived] Anteraper SA, Guell X, Lee YJ, Raya J, Demchenko I, Churchill NW, Frey BN, Hassel S, Lam RW, MacQueen GM, Milev R, Schweizer TA, Strother SC, Whitfield-Gabrieli S, Kennedy SH, Bhat V; CAN-BIND Investigator Team. Cerebello-cerebral Functional Connectivity Networks in Major Depressive Disorder: a CAN-BIND-1 Study Report. Cerebellum. 2023 Feb;22(1):26-36. doi: 10.1007/s12311-021-01353-5. Epub 2022 Jan 13. PMID 35023065
- [Derived] van der Wijk G, Harris JK, Hassel S, Davis AD, Zamyadi M, Arnott SR, Milev R, Lam RW, Frey BN, Hall GB, Muller DJ, Rotzinger S, Kennedy SH, Strother SC, MacQueen GM, Protzner AB. Baseline Functional Connectivity in Resting State Networks Associated with Depression and Remission Status after 16 Weeks of Pharmacotherapy: A CAN-BIND Report. Cereb Cortex. 2022 Mar 4;32(6):1223-1243. doi: 10.1093/cercor/bhab286. PMID 34416758
- [Derived] Suh JS, Fiori LM, Ali M, Harkness KL, Ramonas M, Minuzzi L, Hassel S, Strother SC, Zamyadi M, Arnott SR, Farzan F, Foster JA, Lam RW, MacQueen GM, Milev R, Muller DJ, Parikh SV, Rotzinger S, Sassi RB, Soares CN, Uher R, Kennedy SH, Turecki G, Frey BN. Hypothalamus volume and DNA methylation of stress axis genes in major depressive disorder: A CAN-BIND study report. Psychoneuroendocrinology. 2021 Oct;132:105348. doi: 10.1016/j.psyneuen.2021.105348. Epub 2021 Jun 29. PMID 34229186
- [Derived] Allen TA, Harkness KL, Lam RW, Milev R, Frey BN, Mueller DJ, Uher R, Kennedy SH, Quilty LC. Interactions between neuroticism and stressful life events predict response to pharmacotherapy for major depression: A CAN-BIND 1 report. Personal Ment Health. 2021 Nov;15(4):273-282. doi: 10.1002/pmh.1514. Epub 2021 May 18. PMID 34008342
- [Derived] Morton E, Bhat V, Giacobbe P, Lou W, Michalak EE, McInerney S, Chakrabarty T, Frey BN, Milev RV, Muller DJ, Parikh SV, Rotzinger S, Kennedy SH, Lam RW; CAN-BIND Investigator Team. Predictors of Quality of Life Improvement with Escitalopram and Adjunctive Aripiprazole in Patients with Major Depressive Disorder: A CAN-BIND Study Report. CNS Drugs. 2021 Apr;35(4):439-450. doi: 10.1007/s40263-021-00803-2. Epub 2021 Apr 16. PMID 33860922
- [Derived] Chakrabarty T, McInerney SJ, Torres IJ, Frey BN, Milev RV, Muller DJ, Rotzinger S, Kennedy SH, Lam RW; CAN-BIND Investigator Team. Cognitive Outcomes with Sequential Escitalopram Monotherapy and Adjunctive Aripiprazole Treatment in Major Depressive Disorder: A Canadian Biomarker Integration Network in Depression (CAN-BIND-1) Report. CNS Drugs. 2021 Mar;35(3):291-304. doi: 10.1007/s40263-021-00793-1. Epub 2021 Mar 8. PMID 33683582
- [Derived] Vaccarino AL, Kalali AH, Blier P, Gilbert Evans S, Engelhardt N, Foster JA, Frey BN, Greist JH, Kobak KA, Lam RW, MacQueen G, Milev R, Muller DJ, Parikh SV, Placenza FM, Rizvi SJ, Rotzinger S, Sheehan DV, Sills T, Soares CN, Turecki G, Uher R, Williams JBW, Kennedy SH, Evans KR. THE DEPRESSION INVENTORY DEVELOPMENT SCALE: Assessment of Psychometric Properties Using Classical and Modern Measurement Theory in a CAN-BIND Trial. Innov Clin Neurosci. 2020 Jul 1;17(7-9):30-40. PMID 33520402
- [Derived] Ge R, Hassel S, Arnott SR, Davis AD, Harris JK, Zamyadi M, Milev R, Frey BN, Strother SC, Muller DJ, Rotzinger S, MacQueen GM, Kennedy SH, Lam RW, Vila-Rodriguez F. Structural covariance pattern abnormalities of insula in major depressive disorder: A CAN-BIND study report. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Dec 20;111:110194. doi: 10.1016/j.pnpbp.2020.110194. Epub 2020 Dec 6. PMID 33296696
- [Derived] Uher R, Frey BN, Quilty LC, Rotzinger S, Blier P, Foster JA, Muller DJ, Ravindran AV, Soares CN, Turecki G, Parikh SV, Milev R, MacQueen G, Lam RW, Kennedy SH; CAN-BIND Investigator Team. Symptom Dimension of Interest-Activity Indicates Need for Aripiprazole Augmentation of Escitalopram in Major Depressive Disorder: A CAN-BIND-1 Report. J Clin Psychiatry. 2020 Jun 16;81(4):20m13229. doi: 10.4088/JCP.20m13229. PMID 32558407
- [Derived] Dunlop K, Rizvi SJ, Kennedy SH, Hassel S, Strother SC, Harris JK, Zamyadi M, Arnott SR, Davis AD, Mansouri F, Schulze L, Ceniti AK, Lam RW, Milev R, Rotzinger S, Foster JA, Frey BN, Parikh SV, Soares CN, Uher R, Turecki G, MacQueen GM, Downar J. Clinical, behavioral, and neural measures of reward processing correlate with escitalopram response in depression: a Canadian Biomarker Integration Network in Depression (CAN-BIND-1) Report. Neuropsychopharmacology. 2020 Jul;45(8):1390-1397. doi: 10.1038/s41386-020-0688-x. PMID 32349119
- [Derived] Davis AD, Hassel S, Arnott SR, Harris J, Lam RW, Milev R, Rotzinger S, Zamyadi M, Frey BN, Minuzzi L, Strother SC, MacQueen GM, Kennedy SH, Hall GB. White Matter Indices of Medication Response in Major Depression: A Diffusion Tensor Imaging Study. Biol Psychiatry Cogn Neurosci Neuroimaging. 2019 Oct;4(10):913-924. doi: 10.1016/j.bpsc.2019.05.016. Epub 2019 Jun 12. PMID 31471185
- [Derived] Kennedy SH, Lam RW, Rotzinger S, Milev RV, Blier P, Downar J, Evans KR, Farzan F, Foster JA, Frey BN, Giacobbe P, Hall GB, Harkness KL, Hassel S, Ismail Z, Leri F, McInerney S, MacQueen GM, Minuzzi L, Muller DJ, Parikh SV, Placenza FM, Quilty LC, Ravindran AV, Sassi RB, Soares CN, Strother SC, Turecki G, Vaccarino AL, Vila-Rodriguez F, Yu J, Uher R; CAN-BIND Investigator Team. Symptomatic and Functional Outcomes and Early Prediction of Response to Escitalopram Monotherapy and Sequential Adjunctive Aripiprazole Therapy in Patients With Major Depressive Disorder: A CAN-BIND-1 Report. J Clin Psychiatry. 2019 Feb 5;80(2):18m12202. doi: 10.4088/JCP.18m12202. PMID 30840787
- See also: A news article from the Calgary site promoting the CAN-BIND project. — http://www.albertahealthservices.ca/7297.asp
- See also: CAN-BIND study website — http://www.canbind.ca
- See also: "Treating Depression Takes Too Long" — https://www.youtube.com/watch?v=vtJJgxBToWk